CLINICAL TRIAL: NCT04868851
Title: Mobile Health Biometrics to Enhance Exercise and Physical Activity Adherence in Children and Young People with Diabetes
Brief Title: MHealth Biometrics for Young People with Diabetes
Acronym: MOTIVATE-HfH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Liverpool John Moores University (Other)
Collaborators: Oxford University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MOTIVATE HfH
Record Dates: First submitted 2021-04-22; First posted 2021-05-03 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2023-03

CONDITIONS: Diabetes
Keywords: mobile health technology; physical activity; exercise; exercise prescription/ education; exercise adherence
MeSH Terms: conditions — Diabetes Mellitus; Motor Activity

STUDY DESIGN:
Intervention Model Description: pilot, parallel group, randomised controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Here for Health only (Active Comparator): Patients will complete the Here for Health Healthy Lifestyle intervention designed by the Paediatric Diabetes Dietitians at Oxford University Hospitals NHS Foundation Trust.
  Interventions: Behavioral: Here for Health Only
- mHealth technology assisted exercise counselling (mHealth) (Experimental): Patients will complete the Here for Health Healthy Lifestyle intervention before completing a 12 week mHealth technology assisted exercise counselling intervention. Participants will co-develop a 3-month structured exercise and PA programme, with support from an exercise specialist. All participants will have 5 exercise consultations with their exercise specialist. The intervention will be supported by 3 mHealth elements; 1) a wrist worn fitness watch, 2) a smartphone app for patients, and 3) a coaching website for the exercise specialist. The 3 elements will be synced, allowing data to be transferred between platforms.
  Interventions: Behavioral: mHealth technology assisted exercise counselling

INTERVENTIONS:
Behavioral: Here for Health Only — Patients will complete the Here for Health Healthy Lifestyle intervention designed by the Paediatric Diabetes Dietitians at Oxford University Hospitals NHS Foundation Trust.
  Arms: Here for Health only
Behavioral: mHealth technology assisted exercise counselling — Patients will complete the Here for Health intervention before completing a 3 month exercise and physical activity intervention supported by mHealth technology
  Arms: mHealth technology assisted exercise counselling (mHealth)

SUMMARY:
The investigators aim to undertake a feasibility randomised controlled trial (RCT) to investigate whether mHealth technology, allowing biometric informed feedback and coaching on exercise and PA, can be effective in children with diabetes. The overall objective is to have an evidence-based exercise and PA intervention ready to evaluate in a future RCT.

DETAILED DESCRIPTION:
Staff from the Children's Diabetes team at Oxford University Hospitals NHS Foundation Trust will identify patients during routine multidisciplinary team (MDT) clinics. 30 young people with diabetes will be recruited and randomly assigned to one of two groups (Active control n=15, Intervention n=15). Following baseline measures all patients will then complete the 12 week Here for Health (HfH) Healthy lifestyle programme designed by the Diabetes team at Oxford University Hospitals NHS Foundation Trust. Following the initial HfH intervention period assessments will be repeated (T2) before a second 12 week intervention period is completed. Active control patients will receive no further input. The intervention group will be provided with exercise counselling and to support this they will also be provide with a wristwatch that can monitor everyday activity and their heart rate, a smartphone app and access to a website. The intervention group will also participate in 5 consultations with an exercise specialist to plan their exercise programme and be updated on their progress towards physical activity targets. Weekly text message updates will also provide feedback to the intervention group with participants able to respond to these updates. Following the second intervention period assessments will be repeated for a final time (T3). Testing at baseline and following the 2 interventions will include changes in physical activity, blood pressure, glycaemia control, body composition and diet.

ELIGIBILITY:
Inclusion Criteria:

* Receiving input from the Here for Health Healthy Lifestyle Programme
* Aged 12-18 years
* Diagnosed with type 1 diabetes
* Type 1 diabetes diagnosis more than 1 year ago
* Hypoglycaemic aware or on a continuous glucose monitor (CGM) with alarms
* Willing to attend additional education on managing blood glucose and exercise
* Diagnosed with type 2 diabetes and on a stable metformin dose for 3-months or more
* BMI centile > 91st
* Access to internet-enabled device for video calling

Exclusion Criteria:

* Severe learning/behaviour difficulties
* Severe autism
* Unstable blood glucose levels
* Glucose lowering medications other than metformin
* Underlying medical conditions that contraindicate physical activity

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 18 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Eligibility Rate | Through study completion, an average 32 weeks
  Determine the number of young people referred to the paediatric diabetes team that are eligible to participate
Recruitment rate | Through study completion, an average 32 weeks
  The proportion of eligible patients who would be willing to take part in this trial
Drop out | Through study completion, an average 32 weeks
  Determine the number of young people retained at study completion (i.e., participant drop-out).

SECONDARY OUTCOMES:
Device derived adherence to structured exercise (mHealth technology assisted exercise counselling, Only) | Through study completion, an average 32 weeks
  Number of exercise sessions per week
Device derived duration of exercise (mHealth technology assisted exercise counselling, Only) | Through study completion, an average 32 weeks
  minutes of exercise completed per session
Device derived intensity of structured exercise (mHealth technology assisted exercise counselling, Only) | Through study completion, an average 32 weeks
  intensity of exercise sessions performed (% of HR max)
Device derived physical activity (GENEActiv) | Baseline, the final 2 weeks of intervention period 1 (weeks 10-12), and the final 2 weeks of intervention period 2 (weeks 22-24)
  Minutes of low, moderate and vigorous physical activity
Survey reported exercise behaviour (Godin Leisure Time Exercise Questionnaire (GLTEQ)) | Baseline, 4, 8 12,16, 20, 24 weeks
  Bouts of mild, moderate and strenuous exercise lasting ≥30 minutes
Height | Baseline and immediately following intervention 1 (12 weeks) and 2 (24 weeks)
  Height (m)
Weight | Baseline and immediately following intervention 1 (12 weeks) and 2 (24 weeks)
  Weight (kg)
Body composition | Baseline and immediately following intervention 1 (12 weeks) and 2 (24 weeks)
  bioimpedence (fat mass and lean mass)
Concentration of Hba1c | Baseline and immediately following intervention 1 (12 weeks) and 2 (24 weeks)
  Hba1c
Blood Lipid concentrations | Baseline and immediately following intervention 1 (12 weeks) and 2 (24 weeks)
  Total cholesterol, HDL/LDL, Triglycerides
Glycaemic control | Baseline, immediately following intervention period 1 (12 weeks) and the final 2 weeks of intervention period 2 (weeks 22-24))
  Flash glucose monitoring
Insulin dose | Baseline, immediately following intervention period 1 (12 weeks) and the final 2 weeks of intervention period 2 (weeks 22-24))
  Insulin dose log
Diet | Baseline and immediately following intervention 1 (12 weeks) and 2 (24 weeks)
  Patients will be asked to complete The UK Diabetes and Diet Questionnaire (UKDDQ)
Patient survey on intervention acceptability (mHealth technology assisted exercise counselling) | immediately following intervention 2 (24 weeks)
  Study specific questionnaire
Parent survey on intervention acceptability (mHealth technology assisted exercise counselling) | immediately following intervention 2 (24 weeks)
  Study specific questionnaire
Patient survey on intervention acceptability (Here for Health) | immediately following intervention 1 (12 weeks)
  Study specific questionnaire
Parent survey on intervention acceptability (Here for Health) | immediately following intervention 1 (12 weeks)
  Study specific questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Cocks, PhD, Principal Investigator — Liverpool John Moore University
Locations (2):
- United Kingdom (2):
  - Liverpool John Moores University, Liverpool
  - Oxford University Hospitals NHS Foundation Trust, Oxford

IPD SHARING:
Plan to Share IPD: No
No plan to share